CLINICAL TRIAL: NCT06943508
Title: Effects of Nordic Walk on Balance and Functional Strength in Children With Down Syndrome
Brief Title: Nordic Walk on Balance and Functional Strength in Children With Down Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR/AHS/namra khalid
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Down Syndrome
Keywords: Nordic walking; Balance; Postural Sway; Down Syndrome
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial performed through convenient sampling, in which 32 DS children with age of 8-13 years will be taken randomly after screening and meeting inclusion criteria. Divided into two groups. Control group will recieve conventional therapy for 30 min for 5 days per week. Experimental will recieve nordic walk for 30 min for 5 days per week.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Control: Conventional therapy program for 30 min , 5 days per week during 6 week period
  Interventions: Other: Conventional Therapy
- Group B (Experimental): Experimental: Nordic Walk for 30 min, 5 days per week during 6 week period
  Interventions: Other: Nordic Walk

INTERVENTIONS:
Other: Conventional Therapy — Conventional Therapy group: Group A will be control group which will recieve conventional physical therapy program like curl up, lateral step up and sit to stand for 6 weeks( 5 sessions per week)
  Arms: Group A
Other: Nordic Walk — Nordic Walk group: Group B will recieve Nordic walking for 6 weeks ( 5 sessions per week)
  Arms: Group B

SUMMARY:
Down syndrome (DS) is one of the more commonly occurring genetic disorders, where mental retardation is combined with nutritional diseases. It is caused by having a third copy of chromosome 21, and there exist 3 forms; Simple Trisomy 21, Translocation Trisomy and Mosaic Trisomy. It is coupled with mental retardation, congenital heart defects, gastrointestinal anomalies .Nordic walking exerts beneficial effects on resting heart rate, blood pressure, exercise capacity, maximal oxygen consumption, and quality of life in patients with various diseases and can thus be recommended to a wide range of people as primary and secondary prevention.

This study will aim to examine the effects of Nordic walk on balance and functional strength in children with Down syndrome. A Randomized Controlled Trial will be conducted through convenient sampling 32 subjects will randomly be allocated into two groups. Group A will include 16 children and will receive conventional exercise program.

Group B will include 16 children and will receive Nordic walking program. Each session will be 30 minutes, 5 sessions per week. The total duration of the study will be 6 weeks.

Pediatric berg balance scale and modified time up and go test, and functional strength test will be used as outcome measure Data will be analyzed on SPSS version 29.0, normality of the data will be checked and tests will be applied according to the normality of the data either it will be parametric test or non-parametric based on the normality.

DETAILED DESCRIPTION:
Down syndrome (DS) is one of the more commonly occurring genetic disorders, where mental retardation is combined with nutritional diseases. It is caused by having a third copy of chromosome 21, and there exist 3 forms; Simple Trisomy 21, Translocation Trisomy and Mosaic Trisomy. It is coupled with mental retardation, congenital heart defects, gastrointestinal anomalies, weak neuromuscular tone, dysmorphic features of the head, neck and airways, audio vestibular and visual impairment, characteristic facial and physical features, hematopoietic disorders and a higher incidence of other medical disorders. Children with Down's syndrome (DS) often have greater postural sway and delay in motor development. Muscle weakness and hypotonia, particularly of the lower extremities, are theorized to impair their overall physical health and ability to perform daily activities. Nordic walking exerts beneficial effects on resting heart rate, blood pressure, exercise capacity, maximal oxygen consumption, and quality of life in patients with various diseases and can thus be recommended to a wide range of people as primary and secondary prevention. This study will aim to examine the effects of Nordic walk on balance and functional strength in children with Down syndrome. A Randomized Controlled Trial will be conducted through convenient sampling 32 subjects will randomly be allocated into two groups. Group A will include 16 children and will receive conventional exercise program.

Group B will include 16 children and will receive Nordic walking program. Each session will be 30 minutes, 5 sessions per week. The total duration of the study will be 6 weeks.

Pediatric berg balance scale and modified time up and go test, and functional strength test will be used as outcome measure Data will be analyzed on SPSS version 29.0, normality of the data will be checked and tests will be applied according to the normality of the data either it will be parametric test or non-parametric based on the normality.

ELIGIBILITY:
Inclusion Criteria:

* Children with age group of 8-13

  * Both male and female
  * Functional ability sufficient enough to understand commands, direction and exercise guidance
  * Have ability to walk 60 meters independently according to 6- minute walk test
  * Children who can stand and walk with balance problem as revealed from physical examination having 20 to 42 scores on PBS.

Exclusion Criteria:

Uncontrolled seizures

* Any kind of orthopedic condition
* Registered visually impaired
* Atlanto Axial instability
* Any chest infection

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-05-26 (Estimated)

PRIMARY OUTCOMES:
Pediatric berg balance scale | Baseline, 6th week
  Pediatric balance scale is a modified version of berg balance scale that is used to assess functional balance skills in children. The scale consists of 14 items that are scored from 0 points (lowest function) to 4 points (highest function) with a maximum NORDIC WALK ON BALANCE AND FUNCTIONAL STRENGHT IN CHILDERN WITH DOWN SYNDROME 11 score of 56 points It has good reliability and validity with (ICC=0.997) (r=0.797, p <0.05)
Timed UP & GO (TUG) test | Baseline, 6th week
  The timed UP & GO (TUG) test was developed by Podsiadlo and Richardson in 1991 that is used to assess dynamic balance during the performance of a task. This test measures in second the time required for an individual to stand up from a standard chair with armrest, walk 3m and turn around with reliability and validity of (ICC=0.98; p<0.01)
Functional Strength Test | Baseline, 6th week
  To assess functional performance in children with functional exercises in which the large muscle group that are important for standing and walking are being tested. Three closed kinetic chain exercises were chosen. Subjects were instructed to perform as many repetitions as possible in 30 seconds. ICC value ranged from 0.91 to 0.96

CONTACTS AND LOCATIONS:
Overall Officials: Hafiza Namra Khalid, MS-PPT, Principal Investigator — Study Principal Investigator
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mazurek D, Wyka J. Down syndrome--genetic and nutritional aspects of accompanying disorders. Rocz Panstw Zakl Hig. 2015;66(3):189-94. PMID 26400113